CLINICAL TRIAL: NCT02373046
Title: A Phase 1, Randomized, Single-center, Open-label, 2-sequence, 2-period, Single-dose Crossover Study to Evaluate Bioequivalence (Pharmacokinetics) and to Compare Total 24-hour Urinary Glucose Excretion (Pharmacodynamics) When 400 mg LX4211 is Administered as a Single 400-mg Tablet and 2 × 200-mg Tablets in Healthy Male and Female Subjects
Brief Title: Bioequivalence Study Between 400 mg LX4211 Tablets and 2 X 200 mg LX4211 Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LX4211.1-117-NRM; LX4211.117 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2015-02-16; First posted 2015-02-26 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
MeSH Terms: interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental): 1 × 400-mg LX4211 tablet (fasted conditions)
  Interventions: Drug: LX4211
- Treatment B (Experimental): 2 × 200-mg LX4211 tablets (fasted conditions)
  Interventions: Drug: LX4211

INTERVENTIONS:
Drug: LX4211 — Single dose of LX4211 400 mg as 1 × 400-mg tablet Day 1 or Day 9
Drug: LX4211 — Single dose of LX4211 400 mg as 2 × 200-mg tablets on Day 1 or Day 9

SUMMARY:
This is a randomized, single-center, open-label, 2-sequence, 2-period, single-dose, crossover study to assess the bioequivalence and the total 24-hour urinary glucose excretion (UGE) of 400 mg LX4211 administered as a single 400-mg tablet compared to 2 × 200-mg tablets in healthy subjects under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects ≥18 to ≤55 years of age
* Willing and able to provide written informed consent

Exclusion Criteria:

* Presence of clinically significant physical, laboratory, or ECG findings that, in the opinion of the Investigator and/or Sponsor, may interfere with any aspect of study conduct or interpretation of results
* Existence of any surgical or medical condition that might interfere with the absorption, distribution, metabolism, or excretion of LX4211
* History of renal disease, or significantly abnormal kidney function test at Screening
* History of hepatic disease, or significantly abnormal liver function tests at Screening
* History of any clinically relevant psychiatric, renal, hepatic, pancreatic, endocrine, cardiovascular, neurological, hematological, or GI abnormality

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
AUC | Days 1 to 5, Days 9 to 13
Urinary Glucose Excretion (UGE) | Day 1, Day 9

SECONDARY OUTCOMES:
# of Adverse Events | Day 1-Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, M.D., Study Director — Lexicon Pharmaceuticals, Inc.
Locations (1):
- Lexicon Investigational Site, Dallas, Texas, United States